CLINICAL TRIAL: NCT06813638
Title: Pain Management After Cesarean Section - A Prospective Before-and-After Cohort Study on the Implementation of the Intraoperative Recommendation of the PROSPECT Guidelines
Brief Title: Pain Management After Cesarean Section - A Before-and-After Cohort Study
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Hillerod Hospital, Denmark (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Patricia Duch, Consultant, MD, Nordsjaellands Hospital
Other Study IDs: 102
Record Dates: First submitted 2025-01-20; First posted 2025-02-07 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cesarean Section; Cesarean Delivery; Pain Management; Pain Management in Postoperative Care; Postoperative Pain; Cohort Study; Text Message; Patient Reported Outcome; Wound Infiltration
Keywords: Pain after cesarean; cesarean delivery; cesarean section; postoperative pain; patient reported outcome; Text message; wound infiltration; pain management; cohort
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elective Cesarean Section patients: Our Danish hospital in the Capital Region handles approximately 4,000 births including 400 elective CS annually (Danish birth registry). We evaluate the routinely used protocols in our center before and after modification of the standard protocol. We have a sample size of 100 historical CS patients with prospective data collection from before the implementation. The patients were included in a study testing the feasibility of electronic text messages for questionnaires on pain from December 2022 to June 2023 (Duch). In this study we plan to include elective CS patients after the implementation in a period between January 2025 and April 2025.

SUMMARY:
Inadequate pain relief remains a challenge after Cesarean section (CS) and may significantly impair postoperative recovery. A recent Danish single-center study (n=100) revealed that 66% of elective CS patients experienced severe pain (NRS ≥ 7) during the first 24 hours, with the highest pain scores occurring within the initial 12 hours.

To optimize postoperative pain management for CS patients at the same study center, the investigators have implemented recommendations for pain management from the PROSPECT guideline for procedure-specific postoperative pain management after CS, as recommended by the European Society of Regional Anaesthesia & Pain Therapy.

The study center had already been adhering to the guidelines concerning postoperative care and surgical technique. The investigators have now implemented the second PROSPECT recommendation, focusing on the intraoperative management after delivery, and implemented wound infiltration in combination with an ilio-inguinal field block, before closing the incision after CS, and intravenous dexamethasone (8mg), administered immediately after birth of the baby during CS.

The investigators designed a before-and-after study with the aim of investigating whether the new practice of adding wound infiltration, an ilio-inguinal field block, and intravenous dexamethasone intraoperatively reduces the incidence of postoperative pain in the early period following CS.

DETAILED DESCRIPTION:
Background Inadequate pain relief remains a challenge after Cesarean section (CS) and may significantly impair postoperative recovery. A recent Danish single-center study (n=100) revealed that 66% of elective CS patients experienced severe pain (NRS ≥ 7) during the first 24 hours, with the highest pain scores occurring within the initial 12 hours.

To optimize postoperative pain management for CS patients at the same study center, the investigators have implemented recommendations for pain management from the PROSPECT guideline for procedure-specific postoperative pain management after CS, as recommended by the European Society of Regional Anaesthesia & Pain Therapy.

The PROSPECT guidelines outline four key recommendations for clinical practice: 1) preoperative management, 2) intraoperative management after delivery, 3) postoperative care, and 4) surgical technique (Figure 1).

The study center had already been adhering to the guidelines concerning postoperative care and surgical technique. The investigators have now implemented the second PROSPECT recommendation, focusing on the intraoperative management after delivery, and implemented wound infiltration in combination with an ilio-inguinal field block, before closing the incision after CS.

Studies reports that truncal nerve blocks provide analgesia for between 6 and 12 hours after CS (Hansen). This is particularly relevant in the study center, where patients report the most intense pain during the 6-12 hour period after CS, coinciding with the first mobilization and initiation of breastfeeding.

The investigators have implemented an ilio-inguinal field block, placed using a landmark technique by the surgeon in combination with wound infiltration, at the end of surgery. This technique has demonstrated good pain scores after CS and provides an accessible approach for intraoperative pain management.

Additionally, following the PROSPECT guideline the investigators have implemented intravenous dexamethasone (8mg), administered immediately after birth of the baby during CS. Studies of the CS population show that dexamethasone improves pain scores, prolongs the analgesic effects of local anesthetics, and reduces opioid consumption.

The investigators designed a before-and-after study with the aim of investigating whether the new practice of adding wound infiltration, an ilio-inguinal field block, and intravenous dexamethasone intraoperatively reduces the incidence of postoperative pain in the early period following CS.

Methods Ethics and approvals This study complies with the Helsinki declaration. Participation was voluntary, and informed consent was obtained from each patient during the inclusion process. Consent could be withdrawn at any time. Approval for data collection, handling, and storage re granted by the data protection authority for the Capital Region of Denmark (Region Hovedstaden) with case number P-2023-90. The Research Ethics Committee for the Capital Region of Denmark (Region Hovedstaden) waived the need for approval due to Danish legislation (Case number F-23004686). The study protocol will be available on clinicaltrials.gov.

Study design A prospective, single-center before- and after cohort study. This study evaluates the quality of pain management after CS in the study center following the implementation of intra-operative elements of an established treatment approach (PROSPECT) and is based on patient-reported outcomes and clinical data from electronic health records. The study is not an intervention study. The investigators evaluate the routinely used protocols in the study center before and after modification of the standard protocol.

Setting The study center is a Danish hospital in the Capital Region and handles approximately 4,000 births including 400 elective CS annually (Danish birth registry).

The investigators have a sample size of 100 historical CS patients from the same study center. These patients were included in a study testing the feasibility of electronic text messages for questionnaires on pain from December 2022 to June 2023. In this study the investigators plan to include elective CS patients after the implementation in a period between January 2025 and April 2025.

The setting, eligibility criteria, data collection and prospective collected patient reported outcomes is the same for both groups before and after changing the standard pain management protocol.

Data collection All data are entered directly into the closed and secure system, REDCap. Questionnaires are sent to the patient at 6, 12, 18, 24, and 48 hours after the CS. The questionnaires are delivered to the patient's smartphone as a text message with a link to a questionnaire in REDCap. Time-limits for responses are set at 3 hours after sending questionnaires. Baseline and perioperative data will be extracted from health records.

Development and validation of questions:

The questions for the patient reported outcomes re developed with inspiration from international consensus regarding obstetric recovery, including the incorporation of the Obs-QoR-10 score (Sultan). Patients, maternity staff, anesthetists, and obstetricians was consulted to determine the key areas of focus during the first postoperative days after a cesarean section. Based on this, independent questions were developed and validated by using standardized methods for designing and conducting surveys. The questions were created to be analyzed individually and not to aggregated into a single score. A validated pain score (Numeric rating scale, NRS 0-10) was incorporated to ensure reliability. Subsequently, the questionnaires were programmed in the REDCap database and designed to present well on a smartphone screen. Finally, the questionnaires were set-up to be sent out as a text message via an external server (Sure-SMS, Denmark) with links to the questionnaires in REDCap. The questionnaires consist of 10 short questions that can be answered on the phone in less than three minutes. With an addition of the Obstetric Quality of Recovery questionnaire 24 hours after CS, that consist of 10 short questions.

Anesthesia, surgery, postoperative analgesia, and recovery plan for elective CS At the study center, hyperbaric bupivacaine combined with fentanyl are used for spinal anesthesia for CS. The surgical procedure is performed using the Joel-Cohen method with blunt dissection of tissue layers. The uterus is either repaired extra-abdominally or in situ. Standardized postoperative pain management consist of fixed doses of paracetamol and NSAIDs, supplemented with oral morphine on request. Breastfeeding (if not declined by the mother) are initiated immediately after the birth, either in the operating room or shortly thereafter. Early mobilization within six hours post-CS is encouraged. The urinary catheter is removed after the first mobilization. The general aim for discharge to home are within 48 hours.

The description above indicates that the study center follows the PROSPECT guideline, regarding surgical technique and postoperative pain management as shown in Figure 1 (Box 1 from the PROSPECT guidelines). In addition, the investigators have recently incorporated the PROSPECT recommendations for intraoperative pain management, with intravenous dexamethasone 8 mg administered right after delivery, wound infiltration, and an ilio-inguinal field block.

A total of 40 ml of ropivacaine 3.75 mg/ml is administered as a local anaesthetic for wound infiltration (single shot) and an ilio-inguinal field block, using a landmark technique intended to target areas associated with the iliohypogastric nerve, as well as the anterior rectus muscle fascia, rectus sheath, and subcutaneous tissue).

Participants Patients will be approached for inclusion in the postoperative care unit shortly after the CS and included as continuously as possible in the inclusion period, with the limitation that inclusion will only occur when one of the two site investigators is present at work.

Sample size considerations The sample size estimation was based on the primary outcome: Pain during movement 6 hours after cesarean section (CS), measured using a numeric rating scale (NRS) from 0 to 10. A change of one point on the NRS was deemed clinically relevant. In the "before" group (n = 78), the baseline mean for the primary outcome was NRS 6.76 (SD 1.90). A power analysis performed using G*Power (Faul) with an alpha of 0.05 and a beta of 0.8 indicated that detecting a reduction to NRS 5.76 (SD 1.90) in the "after" group would require a minimum of 45 patients, with an allocation ratio of 2:1.To account for an anticipated non-response rate of approximately 33% for the 6-hour questionnaire, the investigators aim to include 60 patients in the "after" group.

Data Processing and statistics All data will be handled in the secure REDCap database. Descriptive statistics will be used to analyze data. Continuous data will be summarized as median (interquartile range) or mean if the data is normally distributed, and categorical data as frequency (percentage).

To compare the primary and secondary outcomes between the two groups before and after the implementation, the investigators will use a two-sample t-test for continuous variables if the data is normally distributed. For non-normally distributed data, a Wilcoxon rank-sum test will be applied. For categorical variables, a Chi-squared test will be used to compare the distribution of responses between the groups. A p-value of < 0,05 is considered significant.

The investigators will try to minimize missing data as much as possible, by sending questionnaires directly to the participants mobile phones and including the patients face-to-face. The number of missing data will be accounted for when describing data.

All references can be found in the attached protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo planned cesarean section under spinal anesthesia.
* Patients who speak and read Danish and can provide informed consent to participate.
* Patients who have a mobile phone that can receive a text message with a link to a questionnaire that can be accessed on an online website on the phone.
* Age ≥ 18 years

Exclusion criteria:

* The study excludes patients with daily opioid use.
* Multiple pregnancies (gemelli or more).
* Insulin-treated diabetes.
* Chronic pain patients.
* Unplanned CS

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective CS Patients at our center will be approached for inclusion in the postoperative care unit shortly after the CS during the study period
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Pain at movement at 6 hours after Cesarean Section | 6 hours, questionnaire at 6 hours after cesarean section
  Patient reported pain when moving from lying to sitting position, Numeric Rating Scale 0-10, 0=no pain, 10=worst possible pain.

SECONDARY OUTCOMES:
Pain at movement at 12 hours after Cesarean Section | 12 hours, questionnaire at 12 hours after cesarean section
  Patient reported pain when moving from lying to sitting position, Numeric Rating Scale 0-10, 0=no pain, 10=worst possible pain.
Severe pain (NRS ≥ 7) at any time within the first 24 hours after Cesarean Section | 24 hours, questionnaires at 6, 12, 18, 24 hours after cesarean section
  Patient reported pain when moving from lying to sitting position, Numeric Rating Scale 0-10, 0=no pain, 10=worst possible pain.
Opioid consumption during the first 24 hours after CS. (oral morphine equivalents, mg) | 24 hours
  Clinical data from electronic health records, oral morphine equivalents, mg.
Pain at movement at 18 hours after Cesarean Section | 18 hours, questionnaire at 18 hours after cesarean section
  Patient reported pain when moving from lying to sitting position, Numeric Rating Scale 0-10, 0=no pain, 10=worst possible pain.
Pain at movement at 24 hours after Cesarean Section | 24 hours, questionnaire at 24 hours after cesarean section
  Patient reported pain when moving from lying to sitting position, Numeric Rating Scale 0-10, 0=no pain, 10=worst possible pain.
Severe pain (NRS ≥ 7), at any timepoint within the first 24 hours. | 24 hours, questionnaires at 6, 12, 18, 24 hours after cesarean section
  Patient reported pain when moving from lying to sitting position, Numeric Rating Scale 0-10, 0=no pain, 10=worst possible pain.
Pain at rest after Cesarean section. NRS 0-10. | 24 hours, questionnaires at 6, 12, 18, 24 hours after cesarean section
  Patient reported pain at rest, Numeric Rating Scale 0-10, 0=no pain, 10=worst possible pain.
Satisfaction with pain-treatment during the first 24 hours after Cesarean section | 24 hours, questionnaire at 24 hours after cesarean section
  Rated from 0-10; 0=very dissatisfied.10=very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Duch, MD, Principal Investigator — Department of Anaesthesia, University Hospital of Copenhagen, Northern Zealand
Locations (1):
- University Hospital of Copenhagen, Northern Zealand, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All results will be shared in an anonymous form upon reasonable request after the study is published.
Supporting Information: Study Protocol
Time Frame: Data will be collected, analyzed and drafted for publication in 2025.
Access Criteria: The study protocol is uploaded with the registration on Clinical trials 1th February 2025.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT06813638/Prot_SAP_000.pdf